CLINICAL TRIAL: NCT03322826
Title: A Prospective and Multi-center RCT Study of Lymphadenectomy Based on Intraoperative Frozen Pathology for Pulmonary Invasive Adenocarcinoma Presenting With Ground Glass Opacity
Brief Title: Systematic Sampling of Lymph Nodes vs. Lymphadenectomy According to Intraoperative Frozen Pathology for Pulmonary Invasive Adenocarcinoma With Ground-glass Opacity
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai Pulmonary Hospital, Shanghai, China (Other)
Collaborators: Changhai Hospital (Other); Shanghai 10th People's Hospital (Other); Ruijin Hospital (Other); RenJi Hospital (Other)
Responsible Party: Principal Investigator, Chang Chen, Vice President, Shanghai Pulmonary Hospital, Shanghai, China
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SHDC12015116
Record Dates: First submitted 2017-10-23; First posted 2017-10-26 (Actual); Last update posted 2017-12-19 (Actual); Status verified 2017-12

CONDITIONS: Lymph Node Excision
MeSH Terms: interventions — Lymph Node Excision

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Lymphadenectomy (Active Comparator): systematically Lymphadenectomy of the lymph-node stations ATS 2, 4, 7, 8, 9,10,11 on the right side and ATS 5, 6, 7, 8, 9,10,11 on the left side
  Interventions: Procedure: lymphadenectomy
- systematic sampling of the lymph nodes (Experimental): systematic sampling of the lymph-node stations ATS 2, 4, 7, 8, 9,10,11 on the right side and ATS 5, 6, 7, 8, 9,10,11 on the left side
  Interventions: Procedure: systematic sampling of the lymph-node

INTERVENTIONS:
Procedure: systematic sampling of the lymph-node — Systematic Sampling of lymph nodes
  Arms: systematic sampling of the lymph nodes
Procedure: lymphadenectomy — Routine lymph nodes dissection in lung cancer
  Arms: Lymphadenectomy

SUMMARY:
The purpose of this study is to evaluate the impact of systematic sampling of lymph nodes vs. lymphadenectomy on outcome according to intraoperative frozen pathology for pulmonary invasive adenocarcinoma with ground-glass opacity (GGO) after VATS lobectomy.

DETAILED DESCRIPTION:
On HRCT screening, early lung adenocarcinoma often contains a nonsolid component called ground-glass opacity (GGO). In 2011, pulmonary adenocarcinomas were classified into atypical adenomatous hyperplasia (AAH), adenocarcinoma in situ (AIS), minimally invasive carcinoma (MIA) and more extensively invasive adenocarcinoma (IAC) [1]. Early adenocarcinomas with GGO-dominant always mean low-grade malignancy and have an extremely favorable prognosis [2-5]. Previous studies have shown that patients with AAH, AIS and MIA have excellent survival rates (5-year survival rate is approximate 95%) after resection, and only 0.83% - 2.91% patients have lymph node metastasis [6-9]. At present, lymphadenectomy is always undergone in patients with pulmonary adenocarcinoma with ground-glass opacity. However, for MIA patients (especially in T1a-b stage), the appropriate use of lymphadenectomy continues to be debated.

Nowadays, intraoperative frozen pathology is widely used during operation. However, whether sampling of lymph nodes or lymphadenectomy should be performed for GGO lesions according to intraoperative pathological diagnosis is unclear. The aim of this prospective study is to evaluate whether there are any trends regarding the impact of subtypes of invasive adenocarcinoma according to intraoperative frozen pathology in sampling of lymph nodes vs. lymphadenectomy.

ELIGIBILITY:
Inclusion Criteria:

1. A peripheral nodular lesion;
2. The maximum diameters of whole GGO lesions and solid components on lung windows were no more than 3 cm (T1 stage);
3. VATS lobectomy
4. 25%≦Consolidation/Tumor ratio ≦50%
5. ECOG performance status 0-2;
6. Without distant metastasis;
7. Intraoperative frozen pathology confirmed invasive or minimally invasive adenocarcinoma.
8. No operation contraindication
9. Cardiovascular: Cardiac function normal
10. Renal: Creatinine clearance greater than 60 ml/min
11. The expected survival after surgery ≥ 6 months
12. Must be able to sign written informed consent form

Exclusion Criteria:

1. Age less than 18 years old
2. Known hereditary bleeding disorder with history of post-operative hemorrhage
3. Patients maintained on chronic anticoagulation (eg Coumadin therapy)
4. Known hematogenous disorder
5. Known primary or secondary malignancy
6. Pregnant or breast-feeding women;
7. Clinically significant heart disease;
8. Patients who are unwilling or unable to comply with study procedures;
9. Receiving immunosuppressive therapy;
10. HIV/AIDS.
11. Multiple lesions in lung

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 600 (Estimated)
Dates: Start 2017-12-08 (Actual); Primary Completion 2021-10-28 (Estimated); Study Completion 2023-10-28 (Estimated)

PRIMARY OUTCOMES:
recurrence-free survival | five years after surgery
  recurrence-free survival status of patients after surgery

SECONDARY OUTCOMES:
Overall Survival | five years after surgery
  survival status of patients after surgery
Morbidity rate | up to 30 days after surgery
  the rates of complications related to treatment during perioperative period
Mortality rate | up to 30 days after surgery
  the rates of death related to treatment during perioperative period

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Pulmonary Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Tsutani Y, Miyata Y, Nakayama H, Okumura S, Adachi S, Yoshimura M, Okada M. Appropriate sublobar resection choice for ground glass opacity-dominant clinical stage IA lung adenocarcinoma: wedge resection or segmentectomy. Chest. 2014 Jan;145(1):66-71. doi: 10.1378/chest.13-1094. PMID 24551879
- [Result] Ye B, Cheng M, Li W, Ge XX, Geng JF, Feng J, Yang Y, Hu DZ. Predictive factors for lymph node metastasis in clinical stage IA lung adenocarcinoma. Ann Thorac Surg. 2014 Jul;98(1):217-23. doi: 10.1016/j.athoracsur.2014.03.005. Epub 2014 May 17. PMID 24841547